CLINICAL TRIAL: NCT04877548
Title: Randomized Pilot Study to Measure the Effects of an Acute Intake of Fermented Fruits Flours on Postprandial Glycaemic Response and Metabolic Profile
Brief Title: Powdered Fermented Fruits for Glycemia Reduction
Acronym: P2F-GR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL20_1032
Record Dates: First submitted 2021-04-26; First posted 2021-05-07 (Actual); Last update posted 2021-09-20 (Actual); Status verified 2021-09

CONDITIONS: Cardiometabolic Risk Factors; Obesity, Abdominal
Keywords: Postprandial glycaemia; Dietary fibers; Cardiometabolic risk; Fermented fruit flour
MeSH Terms: conditions — Obesity, Abdominal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Fermented orange flour (Experimental): Volunteers will have to consume a standardized breakfast including fermented orange flour and presenting 50g of available carbohydrates
  Interventions: Other: Fermented orange flour
- Fermented grape flour (Experimental): Volunteers will have to consume a standardized breakfast including fermented grape flour and presenting 50g of available carbohydrates
  Interventions: Other: Fermented grape flour
- Control (Placebo Comparator): Volunteers will have to consume a standardized breakfast without fermented flour but also presenting 50g of available carbohydrates
  Interventions: Other: Control

INTERVENTIONS:
Other: Fermented orange flour — Volunteers will have to consume a standardized breakfast including fermented orange flour and presenting 50g of available carbohydrates
  Arms: Fermented orange flour
Other: Fermented grape flour — Volunteers will have to consume a standardized breakfast including fermented grape flour and presenting 50g of available carbohydrates
  Arms: Fermented grape flour
Other: Control — Volunteers will have to consume a standardized breakfast without fermented flour but also presenting 50g of available carbohydrates
  Arms: Control

SUMMARY:
The aim of the study is to evaluate the effects of an acute intake of two fermented fruits flours as part of a standardized breakfast, in comparison with the acute intake of a standardized breakfast without fermented fruits flour but with the same amount of available carbohydrates, on postprandial glycaemic response and overall metabolism in subjects at cardiometabolic risk.

The metabolic parameters will be assessed in fasting and in postprandial period after the consumption of the standardized breakfast.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index between 25 and 35 kg/m2 inclusive
* Waist circumference > 80 cm for women and > 96 cm for men
* Fibers intake ≤ 25g/day

Exclusion Criteria:

* History of digestive surgery or diseases
* Current or recent (<12 weeks) intake of antibiotics or gastro-intestinal medicinal product
* Current probiotics, prebiotics, fibers complement, and/or any products modulating glucose and lipid metabolism
* Volunteer with a dietary restriction (vegetarian or high-protein diet for example)
* Current weight loss diet
* Pregnant or lactating woman or woman who do not use effective contraception
* Drinking more than 3 glasses of alcohol per day (>30g/day)
* Smoking volunteer

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-09-07 (Actual); Primary Completion 2022-08-01 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
Incremental area under curve (iAUC 0-240 min) of postprandial glycaemia in response to an acute intake of different standardized breakfast including or not a fermented fruits flour but which all contain similar amount of available carbohydrate. | Through study completion, an average of 18 days
  Glycaemia will be measured at time t-30, 0, 15, 30, 45, 60, 90, 120, 180, 240 (when taking the standardized breakfast).

SECONDARY OUTCOMES:
Maximum value, total and incremental area under curve (iArea Under Curve and tArea Under Curve 0-120, 0-240 and 120-240 min) of glycaemia and insulinemia | Through study completion, an average of 18 days
  Glycaemia and insulinemia will be measured at time t-30, 0, 15, 30, 45, 60, 90, 120, 180, 240 (when taking the standardized breakfast).
Glycaemia tArea Under Curve/insulinemia tArea Under Curve ratio (0-120 and 0-240 min) | Through study completion, an average of 18 days
  Glycaemia and insulinemia will be measured at time t-30, 0, 15, 30, 45, 60, 90, 120, 180, 240 (when taking the standardized breakfast).
Maximum value, total and incremental area under curve (iArea Under Curve and tArea Under Curve 0-120, 0-240 and 120-240 min) of digestive hormones (GLP-1 and ghrelin) | Through study completion, an average of 18 days
  GLP-1 and ghrelin concentrations will be measured at time t-30, 0, 15, 30, 45, 60, 90, 120, 180, 240 and t0, 60, 120, 180, 240 respectively (when taking the standardized breakfast).
Maximum value, total and incremental area under curve (iArea Under Curve and tArea Under Curve 0-240 min) of expired gases (H2, CH4) | Through study completion, 24 hours following the last day
  Expired gases concentrations will be measured at time t-30, 0, 60, 120, 180, 240, 360, 480, before the diner and the breakfast next day (24 hours following the standardized breakfast intake).
Oxidation of energy substrates (carbohydrates, lipids, proteins) and induced-food thermogenesis | Through study completion, an average of 18 days
  Indirect calorimetry measurement during the postprandial period (0-240 min) (when taking the standardized breakfast).
Satiety and digestive tolerance | Through study completion, 24 hours following the last day
  Visual analogue scales (VAS) on gastrointestinal symptoms and questionnaires on the consistency and frequency of stools completed, when taking the standardized breakfast (24 hours following the standardized breakfast intake).
Baseline characteristics | Day 0 (at fasting before the standardized breakfast intake)
  Anthropometric parameters
  * height (cm),
  * waist and hip circumference (cm),
Dietary intake | Through study completion, an average of 18 days
  Dietary records completed (the day before and the day of the standardized breakfast intake).
Baseline characteristics | Day 0 (at fasting before the standardized breakfast intake)
  Anthropometric parameters:
  - weight (kg)
Baseline characteristics | Day 0 (at fasting before the standardized breakfast intake)
  Anthropometric parameters:
  - body composition (lean body mass and fat mass by impedance)
Baseline characteristics | Day 0 (at fasting before the standardized breakfast intake)
  Metabolic parameters (glycaemia, insulinemia).
Baseline characteristics | Day 0 (at fasting before the standardized breakfast intake)
  Digestive hormones (GLP-1, ghrelin)
Baseline characteristics | Day 0 (at fasting before the standardized breakfast intake)
  Expired gases (H2, CH4)
Baseline characteristics | Day 0 (at fasting before the standardized breakfast intake)
  Resting metabolic rate.

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie FEUGIER-FAVIER, MD, Principal Investigator — Centre de Recherche en Nutrition Humaine Rhône-Alpes
Locations (1):
- Centre de Recherche en Nutrition Humaine Rhône-Alpes, Pierre-Bénite, France